CLINICAL TRIAL: NCT02215629
Title: A Phase I Dose Escalation Study of VS-4718, A Focal Adhesion Kinase Inhibitor, In Subjects With Relapsed or Refractory Acute Myeloid Leukemia or B-Cell Acute Lymphoblastic Leukemia
Brief Title: Dose Escalation Study in Acute Myeloid or B-Cell Acute Lymphoblastic Leukemia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Verastem, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VS-4718-102
Record Dates: First submitted 2014-08-07; First posted 2014-08-13 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2015-10

CONDITIONS: Relapsed or Refractory Acute Myeloid Leukemia; Relapsed or Refractory B-Cell Acute Lymphoblastic Leukemia
Keywords: Leukemia; Acute Leukemia; Relapsed Leukemia; Refractory Leukemia; Acute Myeloid Leukemia; B-Cell Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Recurrence; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Leukemia | interventions — PND 1186

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental VS4718 (Experimental): Oral VS-4718 administered BID during a 28 day cycle.
  Interventions: Drug: VS-4718

INTERVENTIONS:
Drug: VS-4718

SUMMARY:
The main purpose of this study is to test the safety and efficacy of VS-4718 in two types of leukemia patients and to find the right dose of VS-4718 for future clinical trials.

Other purposes of this study include:

* Testing for study drug VS-4718 levels in blood over time and what happens to the study drug in patients.
* To find out if there are certain biomarkers in leukemia patients that predict if and how 4718 study drug may or may not work.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Pathologic confirmation of AML or B-ALL
* Must have relapsed or refractory AML or B-ALL with no alternate therapy of proven benefit
* ECOG status of 0 or 1
* Adequate renal function [creatinine less than or equal to 1.5x ULN] or GFR of at least 60mL/min
* Adequate hepatic function via total bilirubin, AST, and ALT
* Corrected QT interval of less than 470 ms (via Fridericia correction formula)
* Negative pregnancy test for women of child bearing potential
* Willingness to use adequate birth control throughout participation for both men and women

Exclusion Criteria:

* Diagnosis of acute promyelocytic leukemia
* Active grade 2 or higher acute GVHD at time of study entry or active chronic GVHD (moderate or severe)
* Gastrointestinal conditions which could interfere with the swallowing or absorption of study medication
* Diagnosis of currently active CNS leukemia
* Known infection with HIV or AIDS (testing not required)
* Known active Hepatitis A, B or C (testing not required)
* Patients being actively treated for a secondary malignancy
* Cancer-directed therapy within 14 days of the first dose of study drug or 5 half-lives, whichever is longer
* Major surgery within 28 days prior to the first dose of study drug
* Use of an investigational drug within 28 days or 5 half-lives whichever is longer
* Women who are pregnant or breastfeeding
* Evidence of uncontrolled infections requiring antibiotic therapy; potential subjects with known or suspected infections on stable antibiotic therapy for 72 hours may be enrolled
* Uncontrolled intercurrent illness including symptomatic congestive heart failure, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2016-09 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
To find the maximum tolerated dose of VS-4718 | Dose Escalation will occurr according to the standard 3+3 design where three subjects are dosed with the same dosage in the first Cycle (of 28 days); subjects will be evaluated for DLTs on Days: 1, 8, 15, 22 and 28 of first Cycle
  In the absence of a dose limiting toxicity (DLT), each subject will receive VS-4718 for a minimum of 28 days of continuous daily dosing (1 cycle), and may continue to receive additional cycles until disease progression or other treatment discontinuation criteria have been met. It is estimated that subjects could potentially receive VS-4718 for up to an additional 2-3 cycles before withdrawal criteria apply.
Safety and Tolerability of VS-4718 Measurements | Safety and tolerability of VS-4718 will be evaluated in each Cycle of 28 days; more specifically, evaluations will occur at a minimum on Days 1, 8, 15, 22, and 28 of the first Cycle
  Specific key measures/observations used to assess safety and tolerability will be: serious adverse events, incidence and severity of adverse events, physical exams (including vital sign measurements), ECGs, and clinical laboratory evaluations (chemistry, hematology, coagulation, urinalysis)

SECONDARY OUTCOMES:
Measure Pharmacokinetics of VS-4718 | Measured concentrations during Cycle 1 on Days 1, 2, 15, and 16. Also on Cycle 2 Day 1 for subjects that continue on study after Cycle 1.
  Systemic VS-4718 concentration as measured in plasma samples versus time by dosing cohort using descriptive statistics

CONTACTS AND LOCATIONS:
Overall Officials: Hagop Youssoufian, MD, Study Chair — Verastem, Inc.